CLINICAL TRIAL: NCT01151241
Title: Outpatient Versus Inpatient Continuous Brachial Plexus Block for Complex Arthroscopic Elbow Surgery: Safety and Functional Outcome
Brief Title: Early Discharge in Patients Undergoing Elbow Arthroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-0120-A
Record Dates: First submitted 2010-06-24; First posted 2010-06-28 (Estimated); Last update posted 2015-02-24 (Estimated); Status verified 2015-02

CONDITIONS: Elbow Arthroscopy Surgery
Keywords: elbow surgery; infraclavicular nerve block; continuous passive motion; ultrasound guided regional anesthesia; early discharge

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early discharge (Experimental): Patients will be discharged home on the first day after surgery, with infraclavicular catheter infusion of local anesthetic in place.
  Interventions: Procedure: Elbow arthroscopy with infraclavicular nerve block and continuous local anesthetic infusion to day 3 post op.; Other: Early Discharge
- Normal Discharge (Active Comparator): Patients will remain in hospital and be discharged per current discharge criteria, once the infraclavicular catheter has been removed on day 3 post op. Typical discharge occurs on day 3 or 4 post op.
  Interventions: Procedure: Elbow arthroscopy with infraclavicular nerve block and continuous local anesthetic infusion to day 3 post op.; Other: Normal Discharge

INTERVENTIONS:
Procedure: Elbow arthroscopy with infraclavicular nerve block and continuous local anesthetic infusion to day 3 post op. — Patients undergoing elbow arthroscopy surgery will receive standard anesthesia/analgesia, including infraclavicular nerve block and general anesthesia for surgery followed by infraclavicular catheter infusion of local anesthetic until day 3 after surgery.
Other: Early Discharge — Patients will be discharged home on the first day after surgery, with infraclavicular catheter infusion of local anesthetic in place.
  Arms: Early discharge
Other: Normal Discharge — Patients will remain in hospital and be discharged per current discharge criteria, once the infraclavicular catheter has been removed on day 3 post op. Typical discharge occurs on day 3 or 4 post op.
  Arms: Normal Discharge

SUMMARY:
Patients undergoing elbow arthroscopy surgery will receive standard anesthesia and analgesia (infraclavicular nerve block combined with general anesthesia for surgery; continuous infusion via infraclavicular catheter to day 3 post op). Patients in the experimental group will be discharged home after one day, with infraclavicular catheter in place; patients in the comparator group will stay in hospital for 3 or 4 days, per standard practice. The study will compare range of motion as the primary endpoint, in a non-inferiority design, to see if early discharge is feasible while providing similar recovery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective complex arthroscopic elbow surgery requiring postoperative CPM - synovectomy, capsulectomy, extensive debridement, contracture release, osteocapsular arthroplasty.
* ASA I-III

Exclusion Criteria:

* Age>65
* Cognitively challenged patients
* Severe COPD
* Patients who, on their own or with the assistance of a caregiver, are not confident of being able to remove the local anesthetic infusion catheter at home
* Psychiatric history
* Allergy to ropivacaine.
* Opioid tolerance (>60mg oral morphine or equivalent/day)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-07; Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Range of Motion | 1 year
  Range of motion at the elbow will be measured vs. baseline to determine surgical success.

SECONDARY OUTCOMES:
Post-operative analgesia | 3 days
  Pain scores, by visual analogue scale, will be used to determine patient satisfaction with analgesia to day 3 after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Anahi Perlas, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada